CLINICAL TRIAL: NCT05975333
Title: ChronCan (Chronicling Cancer): Piloting a Novel Writing Intervention With Adolescents and Young Adults With Cancer
Brief Title: Writing Intervention With Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ChronCan; NCI-2023-06074 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cancer Patients; Communication Research
Keywords: Adolescents; Young Adults; Writing Intervention; Interview
MeSH Terms: interventions — Functional Laterality; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Adolescents and young adults (AYA) patients aged 15-25 years currently receiving cancer-directed therapy at St. Jude Children's Research Hospital
  Interventions: Behavioral: Writing; Behavioral: Interview

INTERVENTIONS:
Behavioral: Writing — Participants will be asked to write about their experiences with cancer, guided by several specific open-ended writing prompts to spark ideas.
Behavioral: Interview — Following completion of the writing exercise, participants will reflect on their experiences with the writing intervention in a semi-structured private interview with a member of the research team.
  Other Names: Questions

SUMMARY:
Young people with cancer have difficult experiences and writing exercises may help improve their well-being. However, very few studies have examined how a creative writing activity might be useful for young people with cancer. In this pilot study, researchers at St. Jude Children's Research Hospital hope to explore whether teenagers and young adults with cancer want to participate in a writing exercise and whether they find it to be valuable.

Primary Objective

To assess the feasibility and acceptability of a writing-based narrative medicine intervention for adolescent and young adult patients with cancer.

DETAILED DESCRIPTION:
Participants will be given the opportunity to write about their experiences with cancer, with support and guidance from an expert writer. Participants will meet briefly with the expert at the start of the exercise (15-30 minutes), and they can choose to meet 1-3 additional times with the expert over the next 2 months to receive further support if they wish.

After completing the writing exercise, participants will do an informal interview to share their thoughts about whether the experience of writing felt helpful or not. The post-intervention interview will occur at around 2 months after enrollment, +/- 1 month. Patients may participate in a second informal semi-structured interview 6 to 12 months after completing the first interview. Additionally, bereaved parents may participate in an informal interview on study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-25
* Currently receiving cancer-directed therapy
* Active patient at St. Jude Children's Research Hospital
* Parent of a ChronCan participant who has passed away

Exclusion Criteria:

* Does not meet the inclusion criteria
* If the parents have not responded or not interviewed till December 31, 2025.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of touchpoints that participants have with the narrative medicine expert/guide | During the narrative exercise, up to 2 months after enrollment
  To determine intervention feasibility, the number of touchpoints that participants have with the narrative medicine expert/guide will be tracked
Number of participants who complete the writing exercise | During the narrative exercise, up to 2 months after enrollment
  To determine intervention feasibility, the number of participants who complete the writing exercise will be tracked
Intervention acceptability | Post-intervention interview will occur after the narrative exercise is completed at around 2 months after enrollment, +/- 1 month
  Comparison of acceptability between participants who did/did not participate in the optional check-ins. Analysis of de-identified semi-structured interviews will be done. Interviews will be recorded, transcribed, de-identified, and analyzed using content analysis, an inductive approach that includes memo-writing, codebook development, coding, reconciliation, and synthesis to identify emerging patterns and themes.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Kaye, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT05975333/ICF_000.pdf